CLINICAL TRIAL: NCT03272737
Title: Effect of Low Intensity Strength Training Combined With Moderate Blood Flow Restriction on Muscle Vasodilatation and Arterial Stiffness in Elders With Low Gait Velocity.
Brief Title: Low Intensity Training Combined With KAATSU on Muscle Vasodilatation and Arterial Stiffness in the Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/07993-3
Record Dates: First submitted 2017-07-11; First posted 2017-09-06 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2020-03

CONDITIONS: Frail Elderly Syndrome
Keywords: KAATSU; Cardiovascular system; Elderly

STUDY DESIGN:
Intervention Model Description: Group 1: Blood flow restriction + low intensity strength exercise Group 2: Low intensity strength exercise
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Traditional strength exercise (Active Comparator): This group will be carried out to knee extension exercise without blood flow restriction.
  Interventions:
  * Plethysmography;
  * Protocols of isometric exercise;
  * Pulse wave Velocity (PWV);
  * Flow-mediated dilatation (FMD);
  * Arterial pressure and blood pressure;
  * Quality of life (Euro Qol);
  * 1RM test
  * Speed gait test
  * Anthropometric Assessment
  Interventions: Procedure: 1RM Test; Procedure: Speed gait test; Device: Venous occlusion plethysmography protocol; Device: Measurement of Arterial Stiffness - Pulse Wave Analysis and Velocity; Device: Isometric handgrip exercise protocol; Device: Vasodilatory capacity; Device: Basal blood flow and vasodilatory capacity - Flow mediated dilation (FMD); Diagnostic Test: Quality of Life EuroQol-5 Domain; Other: Anthropometric Assessment
- Strength exercise with KAATSU (Active Comparator): This group will be carried out to knee extension exercise with partial blood flow restriction.
  Interventions:
  * Plethysmography;
  * Protocols of isometric exercise;
  * Pulse wave Velocity (PWV);
  * Flow-mediated dilatation (FMD);
  * Arterial pressure and blood pressure;
  * Quality of life (Euro Qol);
  * 1RM test
  * Speed gait test
  * Anthropometric Assessment
  Interventions: Procedure: 1RM Test; Procedure: Speed gait test; Device: Venous occlusion plethysmography protocol; Device: Measurement of Arterial Stiffness - Pulse Wave Analysis and Velocity; Device: Isometric handgrip exercise protocol; Device: Vasodilatory capacity; Device: Basal blood flow and vasodilatory capacity - Flow mediated dilation (FMD); Diagnostic Test: Quality of Life EuroQol-5 Domain; Other: Anthropometric Assessment

INTERVENTIONS:
Procedure: 1RM Test — The dynamic force of the lower limb muscles will be evaluated by the maximal repetition of knee extension and leg press exercise, according to the protocol presented in a previous study [37]. The elderly will perform a warm up consisting of 1 series with 10 unloaded repetitions. After the warm up, the mass to be lifted will be progressively increased until the maximum load that can be lifted is reached, with a maximum limit of 5 attempts and a 3 to 5 minutes interval between them. The test will be conducted by a physical education professional who will verbally encourage participants throughout these steps and perform the load adjustment at week 5 and 10 (Radaelli, 2014).
  Other Names: 1RM Test (Knee extension and Seated leg press)
Procedure: Speed gait test — To measure the gait speed of participants they will walk 4.6 metres and the time needed to cover this distance is measured. The mean of three attempts is recorded and divided by the distance. The participants included must achieve in the walking test an average of < 0.,9 m/s (Guralnik, 1994).
Device: Venous occlusion plethysmography protocol — A mercury-filled silastic tube, connected to a low-pressure transducer and a plethysmograph (D.E. Hokanson), will be placed around the largest circumference of the calf region. One cuff will be placed around the ankle and another around the thigh. The ankle cuff will be inflated to a supra-systolic pressure 30 seconds before starting the measurements. At 15-second intervals, the cuff around the thigh will be inflated above the venous pressure for a period of seven to eight seconds. Increased tension in the silastic tube reflects an increase in leg volume and vasodilation. The signal of the muscle blood flow wave will be recorded on a polygraph and analysed every minute, averaging three records per minute. The protocol will be performed during 5 minutes of rest, 3 minutes isometric exercise and 2 minutes of recovery (Bahia, 2006).
Device: Measurement of Arterial Stiffness - Pulse Wave Analysis and Velocity — Arterial stiffness will be estimated from the carotid-femoral aortic pulse wave velocity [33]. Carotid-femoral aortic pulse waves will be recorded by tonometry (SphygmoCor, AtCor Medical, Australia). At the same time, an electrocardiogram will be obtained to calculate the wave transit time. Two distances will be measured: the recording point of the carotid artery and the sternal furcula (distance 1) and the sternal furcula and the recording point in the femoral artery (distance 2). The distance travelled by the pulse wave will be calculated as "distance 2" - "distance 1". The carotid-femoral aortic pulse wave velocity will be calculated as: carotid-femoral aortic pulse wave velocity = ¼ * distance travelled by the pulse wave (m) / transit time(s).
Device: Isometric handgrip exercise protocol — In a supine position, the maximal voluntary handgrip force will be determined as the highest force in 3 consecutive attempts using a Jamar hydraulic palmar dynamometer (Asimow Engineering, CAL, USA). For activation of the central command, mechanoreceptors and muscular metaboreceptors the individual will perform, after 5 minutes of rest (baseline records), 3 minutes of exercise at 30% MVC. This manoeuvre isolates the activation of muscle metaboreceptors, observing the selective activation of these. After the isometric handgrip exercise, 2 minutes of recovery will be performed. Throughout the protocol muscle blood flow, blood pressure and heart rate will be recorded.
Device: Vasodilatory capacity — The vasodilatory capacity will be calculated as the percentage of increase of the diameter of the brachial artery and femoral post occlusion in relation to its basal values.
Device: Basal blood flow and vasodilatory capacity - Flow mediated dilation (FMD) — Images of the brachial artery will be recorded by a two-dimensional ultrasonography device with a spectral Doppler and linear transducer (Ultra-0122, Philips, The Netherlands).
Diagnostic Test: Quality of Life EuroQol-5 Domain — This questionnaire is used to estimate the quality of life in participants before and after the study.
Other: Anthropometric Assessment — Anthropometric measurements will be made before and after the training program following the standardization of the International Society for Anthropometric Assessments. The body mass will be measured with an accuracy of 0.1 kg (Filizola). The stature will be obtained by means of the stadiometer with an accuracy of 0.5 cm. The BMI will be calculated as body mass divided by height squared. The circumference of the quadriceps will be measured with a tape measure (Seca) with a precision of 0.1 cm.

SUMMARY:
The purpose of the present study is to evaluate the acute and chronic effect of low intensity strength training with or without moderate blood flow restriction on muscle vasodilation and arterial stiffness in elders with low gait speed. In addition, the responses of prothrombotic factors in blood coagulation, the impact on heart rate and arterial pressure will be assessed.

DETAILED DESCRIPTION:
The investigators propose a study of 26 sedentary elders with low speed gait, supervised by the Hospital Israelita Albert Einstein - Vila Mariana ambulatory. This will be an open clinical trial, prospective, single center, randomized and controlled study. It will be divided into two parts: acute and chronic phases. After signing an informed consent, the participants will be separated in two groups:

Group 1. Resistance exercise with low intensity combined with partial blood flow restriction Group 2. Conventional resistance exercise with low intensity

All of participants will be submitted to interventions tests before and after the period of training which are:

1. Laboratory Tests: Blood tests
2. Plethysmography
3. Handgrip
4. Quality of life questionaire
5. FMD tests
6. Vasodilation capacity

ELIGIBILITY:
Inclusion Criteria:

* Elderly people aged 60 to 85 years, with walking speed <0.8m / s (Guralnik, 1994).

Exclusion Criteria:

* Elderly patients with uncontrolled diabetes mellitus or peripheral neuropathy;
* Symptomatic peripheral obstructive arterial disease or brachial ankle index <0.9;
* Uncontrolled arterial hypertension (BP> 160 / 100mmHg);
* Uncontrolled dyslipidemia (total colostrum> 220mg / dL);
* Infectious with less than 1 month;
* Osteoarticular or neurological problems that prevent training;
* History of anemia, cerebrovascular disease, myocardial infarction in the last 6 months;
* Pior deep venous thrombosis;
* Use of oral anticoagulant;
* Smoking <6 months;
* Use of antiplatelet agents and anticoagulants;
* Cognitive dysfunctions: Mini-mental <24. (Brucki, 2003).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-02-04 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Anthropometric Assessment | Before and after 12 weeksof training
  The body weight will be evaluated using the Filizola brand scale, with an accuracy of 0.1 kg. The stature will be obtained by means of the stadiometer coupled to the Filizola scale, with an accuracy of 0.5 cm. The BMI will be calculated from the weight ratio by height squared. For measures of circumference of the quadriceps, a tape measure of the brand Seca, with precision of 0.1 cm will be used. Anthropometric measurements will be made following the standardization of the International Society for Anthropometric Assessments (ISAK, 2001).

SECONDARY OUTCOMES:
Coagulation factors | Before and after 12 weeksof training
  Blood tests (fibrinogen, Factor VIII, von Willebrand Factor, D-dimer, t-PA and PAI 1)
Tolerability, adherence and adverse effects | Before and after 12 weeks of training
  Evaluate the tolerability, adherence and adverse effects of both groups - Questionnaire
Arterial pressure and heart rate | Before and after 12 weeks of training
  Blood pressure and heart rate measurements
Speed Gait | Before and after 12 weeks of training
  The gait velocity analysis will be performed with time marking, in thousandths of a second, from the displacement of the elderly in a 4.6-meter straight course, based on the measurement (speed / distance traveled).

OTHER OUTCOMES:
Plesthysmography | Before and after 12 weeks of training
  Evaluation of muscle blood flow by plethysmography of venous occlusion
Pulse wave velocity | Before and after 12 weeks of training
  The estimation of the arterial stiffness will be made from the evaluation of the carotid-femoral aortic pulse wave velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana D Janot, Phd, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Instituto Israelita de Ensino e Pesquisa Albert Einstein 's (IIEP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willoughby, D.S. American College of Sports Medicine. ACSM current comment: Resistance Training and the Older Adult. 2012.
- [Result] Amano S, Ludin AF, Clift R, Nakazawa M, Law TD, Rush LJ, Manini TM, Thomas JS, Russ DW, Clark BC. Effectiveness of blood flow restricted exercise compared with standard exercise in patients with recurrent low back pain: study protocol for a randomized controlled trial. Trials. 2016 Feb 12;17:81. doi: 10.1186/s13063-016-1214-7. PMID 26867541
- [Result] Bahia L, de Aguiar LG, Villela NR, Bottino D, Bouskela E. [The endothelium in the metabolic syndrome]. Arq Bras Endocrinol Metabol. 2006 Apr;50(2):291-303. doi: 10.1590/s0004-27302006000200015. Epub 2006 May 23. Portuguese. PMID 16767295
- [Result] Brucki SM, Nitrini R, Caramelli P, Bertolucci PH, Okamoto IH. [Suggestions for utilization of the mini-mental state examination in Brazil]. Arq Neuropsiquiatr. 2003 Sep;61(3B):777-81. doi: 10.1590/s0004-282x2003000500014. Epub 2003 Oct 28. Portuguese. PMID 14595482
- [Result] Cadore EL, Rodriguez-Manas L, Sinclair A, Izquierdo M. Effects of different exercise interventions on risk of falls, gait ability, and balance in physically frail older adults: a systematic review. Rejuvenation Res. 2013 Apr;16(2):105-14. doi: 10.1089/rej.2012.1397. PMID 23327448
- [Result] Cavalcante JL, Lima JA, Redheuil A, Al-Mallah MH. Aortic stiffness: current understanding and future directions. J Am Coll Cardiol. 2011 Apr 5;57(14):1511-22. doi: 10.1016/j.jacc.2010.12.017. PMID 21453829
- [Result] Chen X, Mao G, Leng SX. Frailty syndrome: an overview. Clin Interv Aging. 2014 Mar 19;9:433-41. doi: 10.2147/CIA.S45300. eCollection 2014. PMID 24672230
- [Result] Crenshaw AG, Hargens AR, Gershuni DH, Rydevik B. Wide tourniquet cuffs more effective at lower inflation pressures. Acta Orthop Scand. 1988 Aug;59(4):447-51. doi: 10.3109/17453678809149401. PMID 3421083
- [Result] D'Antona G, Pellegrino MA, Adami R, Rossi R, Carlizzi CN, Canepari M, Saltin B, Bottinelli R. The effect of ageing and immobilization on structure and function of human skeletal muscle fibres. J Physiol. 2003 Oct 15;552(Pt 2):499-511. doi: 10.1113/jphysiol.2003.046276. PMID 14561832
- [Result] Dobrosielski DA, Greenway FL, Welsh DA, Jazwinski SM, Welsch MA; Louisiana Healthy Aging Study. Modification of vascular function after handgrip exercise training in 73- to 90-yr-old men. Med Sci Sports Exerc. 2009 Jul;41(7):1429-35. doi: 10.1249/MSS.0b013e318199bef4. PMID 19516158
- [Result] Esmon CT. Basic mechanisms and pathogenesis of venous thrombosis. Blood Rev. 2009 Sep;23(5):225-9. doi: 10.1016/j.blre.2009.07.002. PMID 19683659
- [Result] Fahs CA, Rossow LM, Thiebaud RS, Loenneke JP, Kim D, Abe T, Beck TW, Feeback DL, Bemben DA, Bemben MG. Vascular adaptations to low-load resistance training with and without blood flow restriction. Eur J Appl Physiol. 2014 Apr;114(4):715-24. doi: 10.1007/s00421-013-2808-3. Epub 2013 Dec 31. PMID 24375201
- [Result] Fielding RA, Rejeski WJ, Blair S, Church T, Espeland MA, Gill TM, Guralnik JM, Hsu FC, Katula J, King AC, Kritchevsky SB, McDermott MM, Miller ME, Nayfield S, Newman AB, Williamson JD, Bonds D, Romashkan S, Hadley E, Pahor M; LIFE Research Group. The Lifestyle Interventions and Independence for Elders Study: design and methods. J Gerontol A Biol Sci Med Sci. 2011 Nov;66(11):1226-37. doi: 10.1093/gerona/glr123. Epub 2011 Aug 8. PMID 21825283
- [Result] Fried LP, Carlson MC, Freedman M, Frick KD, Glass TA, Hill J, McGill S, Rebok GW, Seeman T, Tielsch J, Wasik BA, Zeger S. A social model for health promotion for an aging population: initial evidence on the Experience Corps model. J Urban Health. 2004 Mar;81(1):64-78. doi: 10.1093/jurban/jth094. PMID 15047786
- [Result] Fry CS, Glynn EL, Drummond MJ, Timmerman KL, Fujita S, Abe T, Dhanani S, Volpi E, Rasmussen BB. Blood flow restriction exercise stimulates mTORC1 signaling and muscle protein synthesis in older men. J Appl Physiol (1985). 2010 May;108(5):1199-209. doi: 10.1152/japplphysiol.01266.2009. Epub 2010 Feb 11. PMID 20150565
- [Result] Frontera WR, Suh D, Krivickas LS, Hughes VA, Goldstein R, Roubenoff R. Skeletal muscle fiber quality in older men and women. Am J Physiol Cell Physiol. 2000 Sep;279(3):C611-8. doi: 10.1152/ajpcell.2000.279.3.C611. PMID 10942711
- [Result] Fujimoto N, Prasad A, Hastings JL, Arbab-Zadeh A, Bhella PS, Shibata S, Palmer D, Levine BD. Cardiovascular effects of 1 year of progressive and vigorous exercise training in previously sedentary individuals older than 65 years of age. Circulation. 2010 Nov 2;122(18):1797-805. doi: 10.1161/CIRCULATIONAHA.110.973784. Epub 2010 Oct 18. PMID 20956204
- [Result] Gates PE, Tanaka H, Graves J, Seals DR. Left ventricular structure and diastolic function with human ageing. Relation to habitual exercise and arterial stiffness. Eur Heart J. 2003 Dec;24(24):2213-20. doi: 10.1016/j.ehj.2003.09.026. PMID 14659773
- [Result] Golbidi S, Laher I. Exercise and the aging endothelium. J Diabetes Res. 2013;2013:789607. doi: 10.1155/2013/789607. Epub 2013 Aug 1. PMID 23984434
- [Result] Graham B, Breault MJ, McEwen JA, McGraw RW. Occlusion of arterial flow in the extremities at subsystolic pressures through the use of wide tourniquet cuffs. Clin Orthop Relat Res. 1993 Jan;(286):257-61. PMID 8425355
- [Result] Harris RA, Nishiyama SK, Wray DW, Richardson RS. Ultrasound assessment of flow-mediated dilation. Hypertension. 2010 May;55(5):1075-85. doi: 10.1161/HYPERTENSIONAHA.110.150821. Epub 2010 Mar 29. PMID 20351340
- [Result] Horiuchi M, Okita K. Blood flow restricted exercise and vascular function. Int J Vasc Med. 2012;2012:543218. doi: 10.1155/2012/543218. Epub 2012 Oct 22. PMID 23133756
- [Result] Karabulut M, Sherk VD, Bemben DA, Bemben MG. Inflammation marker, damage marker and anabolic hormone responses to resistance training with vascular restriction in older males. Clin Physiol Funct Imaging. 2013 Sep;33(5):393-9. doi: 10.1111/cpf.12044. Epub 2013 Apr 23. PMID 23701309
- [Result] Kovacic JC, Moreno P, Nabel EG, Hachinski V, Fuster V. Cellular senescence, vascular disease, and aging: part 2 of a 2-part review: clinical vascular disease in the elderly. Circulation. 2011 May 3;123(17):1900-10. doi: 10.1161/CIRCULATIONAHA.110.009118. No abstract available. PMID 21537006
- [Result] Zembron-Lacny A, Dziubek W, Rogowski L, Skorupka E, Dabrowska G. Sarcopenia: monitoring, molecular mechanisms, and physical intervention. Physiol Res. 2014;63(6):683-91. doi: 10.33549/physiolres.932692. Epub 2014 Aug 26. PMID 25157651
- [Result] Lexell J. Human aging, muscle mass, and fiber type composition. J Gerontol A Biol Sci Med Sci. 1995 Nov;50 Spec No:11-6. doi: 10.1093/gerona/50a.special_issue.11. PMID 7493202
- [Result] Libardi CA, Chacon-Mikahil MP, Cavaglieri CR, Tricoli V, Roschel H, Vechin FC, Conceicao MS, Ugrinowitsch C. Effect of concurrent training with blood flow restriction in the elderly. Int J Sports Med. 2015 May;36(5):395-9. doi: 10.1055/s-0034-1390496. Epub 2015 Feb 20. PMID 25700103
- [Result] Loenneke JP, Fahs CA, Rossow LM, Thiebaud RS, Mattocks KT, Abe T, Bemben MG. Blood flow restriction pressure recommendations: a tale of two cuffs. Front Physiol. 2013 Sep 10;4:249. doi: 10.3389/fphys.2013.00249. eCollection 2013. No abstract available. PMID 24058346
- [Result] Manini TM, Yarrow JF, Buford TW, Clark BC, Conover CF, Borst SE. Growth hormone responses to acute resistance exercise with vascular restriction in young and old men. Growth Horm IGF Res. 2012 Oct;22(5):167-72. doi: 10.1016/j.ghir.2012.05.002. Epub 2012 Jun 23. PMID 22727808
- [Result] Manini TM, Visser M, Won-Park S, Patel KV, Strotmeyer ES, Chen H, Goodpaster B, De Rekeneire N, Newman AB, Simonsick EM, Kritchevsky SB, Ryder K, Schwartz AV, Harris TB. Knee extension strength cutpoints for maintaining mobility. J Am Geriatr Soc. 2007 Mar;55(3):451-7. doi: 10.1111/j.1532-5415.2007.01087.x. PMID 17341251
- [Result] Mattar MA, Gualano B, Perandini LA, Shinjo SK, Lima FR, Sa-Pinto AL, Roschel H. Safety and possible effects of low-intensity resistance training associated with partial blood flow restriction in polymyositis and dermatomyositis. Arthritis Res Ther. 2014 Oct 25;16(5):473. doi: 10.1186/s13075-014-0473-5. PMID 25344395
- [Result] Miljkovic N, Lim JY, Miljkovic I, Frontera WR. Aging of skeletal muscle fibers. Ann Rehabil Med. 2015 Apr;39(2):155-62. doi: 10.5535/arm.2015.39.2.155. Epub 2015 Apr 24. PMID 25932410
- [Result] de Souza ER, Correia BS. [Construction of indicators for assessing the policy of reducing accidents and violence for the elderly care]. Cien Saude Colet. 2010 Sep;15(6):2753-62. doi: 10.1590/s1413-81232010000600013. Portuguese. PMID 20922284
- [Result] Moore A, Mangoni AA, Lyons D, Jackson SH. The cardiovascular system. Br J Clin Pharmacol. 2003 Sep;56(3):254-60. doi: 10.1046/j.0306-5251.2003.01876.x. PMID 12919173
- [Result] Nakajima, T. et al. Effects of Exercise and Anti-Aging. Anti-Aging Medicine. 2011. v. 7 n. 8. p. 92-102.
- [Result] Nakajima, T. et al. Effects of low intensity Kaatsu resistance training on skeletal muscle size/strength and endurance capacity in patients with ischemic heart diseases. International Journal of Kaatsu Training Research. 2010. v. 6. p. 1-7.
- [Result] Nakajima, T. et al. Use and safety of KAATSU training; Results of a national survey. International Journal of Kaatsu Training Research. 2006. v. 2. p. 5-13
- [Result] Nazari-Shafti TZ, Cooke JP. Telomerase Therapy to Reverse Cardiovascular Senescence. Methodist Debakey Cardiovasc J. 2015 Jul-Sep;11(3):172-5. doi: 10.14797/mdcj-11-3-172. PMID 26634025
- [Result] Norton K.; Olds T. International Standards for Anthropometric Assessment. 1a ed. Austrália: The International Society for the Advancement of Kinanthropometry; 1996.
- [Result] Odden MC, Peralta CA, Haan MN, Covinsky KE. Rethinking the association of high blood pressure with mortality in elderly adults: the impact of frailty. Arch Intern Med. 2012 Aug 13;172(15):1162-8. doi: 10.1001/archinternmed.2012.2555. PMID 22801930
- [Result] Ozaki H, Loenneke JP, Thiebaud RS, Stager JM, Abe T. Possibility of leg muscle hypertrophy by ambulation in older adults: a brief review. Clin Interv Aging. 2013;8:369-75. doi: 10.2147/CIA.S43837. Epub 2013 Mar 31. PMID 23573066
- [Result] Park DC, Yeo SG. Aging. Korean J Audiol. 2013 Sep;17(2):39-44. doi: 10.7874/kja.2013.17.2.39. Epub 2013 Sep 24. PMID 24653904
- [Result] Park SY, Kwak YS, Harveson A, Weavil JC, Seo KE. Low intensity resistance exercise training with blood flow restriction: insight into cardiovascular function, and skeletal muscle hypertrophy in humans. Korean J Physiol Pharmacol. 2015 May;19(3):191-6. doi: 10.4196/kjpp.2015.19.3.191. Epub 2015 Apr 30. PMID 25954122
- [Result] Radaelli R, Botton CE, Wilhelm EN, Bottaro M, Brown LE, Lacerda F, Gaya A, Moraes K, Peruzzolo A, Pinto RS. Time course of low- and high-volume strength training on neuromuscular adaptations and muscle quality in older women. Age (Dordr). 2014 Apr;36(2):881-92. doi: 10.1007/s11357-013-9611-2. Epub 2014 Jan 11. PMID 24414336
- [Result] Martinez-Ramirez A, Martinikorena I, Gomez M, Lecumberri P, Millor N, Rodriguez-Manas L, Garcia Garcia FJ, Izquierdo M. Frailty assessment based on trunk kinematic parameters during walking. J Neuroeng Rehabil. 2015 May 24;12:48. doi: 10.1186/s12984-015-0040-6. PMID 26003560
- [Result] Ray CA, Rea RF, Clary MP, Mark AL. Muscle sympathetic nerve responses to dynamic one-legged exercise: effect of body posture. Am J Physiol. 1993 Jan;264(1 Pt 2):H1-7. doi: 10.1152/ajpheart.1993.264.1.H1. PMID 8430836
- [Result] Ribeiro, F.A et al. Síndrome metabólica: complacência arterial e a velocidade de onda de pulso. Revista da AMRIGS. 2012. v. 56. n. 1. p. 75-80.
- [Result] Ricci NA, Pessoa GS, Ferriolli E, Dias RC, Perracini MR. Frailty and cardiovascular risk in community-dwelling elderly: a population-based study. Clin Interv Aging. 2014 Oct 6;9:1677-85. doi: 10.2147/CIA.S68642. eCollection 2014. PMID 25336932
- [Result] Russ DW, Grandy JS, Toma K, Ward CW. Ageing, but not yet senescent, rats exhibit reduced muscle quality and sarcoplasmic reticulum function. Acta Physiol (Oxf). 2011 Mar;201(3):391-403. doi: 10.1111/j.1748-1716.2010.02191.x. Epub 2010 Nov 9. PMID 20874807
- [Result] Satoh, I. Kaatsu Training: Application to Metabolic Syndrome. 2011. International Journal of Kaatsu Training Research. 2011. v. 7. p. 7-12.
- [Result] Raskob GE, Angchaisuksiri P, Blanco AN, Buller H, Gallus A, Hunt BJ, Hylek EM, Kakkar A, Konstantinides SV, McCumber M, Ozaki Y, Wendelboe A, Weitz JI; ISTH Steering Committee for World Thrombosis Day. Thrombosis: a major contributor to global disease burden. Arterioscler Thromb Vasc Biol. 2014 Nov;34(11):2363-71. doi: 10.1161/ATVBAHA.114.304488. PMID 25304324
- [Result] Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Blood flow restricted exercise for athletes: A review of available evidence. J Sci Med Sport. 2016 May;19(5):360-7. doi: 10.1016/j.jsams.2015.04.014. Epub 2015 May 9. PMID 26118847
- [Result] Singh M, Stewart R, White H. Importance of frailty in patients with cardiovascular disease. Eur Heart J. 2014 Jul;35(26):1726-31. doi: 10.1093/eurheartj/ehu197. Epub 2014 May 26. PMID 24864078
- [Result] Takarada Y, Takazawa H, Sato Y, Takebayashi S, Tanaka Y, Ishii N. Effects of resistance exercise combined with moderate vascular occlusion on muscular function in humans. J Appl Physiol (1985). 2000 Jun;88(6):2097-106. doi: 10.1152/jappl.2000.88.6.2097. PMID 10846023
- [Result] Thijssen DH, Black MA, Pyke KE, Padilla J, Atkinson G, Harris RA, Parker B, Widlansky ME, Tschakovsky ME, Green DJ. Assessment of flow-mediated dilation in humans: a methodological and physiological guideline. Am J Physiol Heart Circ Physiol. 2011 Jan;300(1):H2-12. doi: 10.1152/ajpheart.00471.2010. Epub 2010 Oct 15. PMID 20952670
- [Result] Verdijk LB, Koopman R, Schaart G, Meijer K, Savelberg HH, van Loon LJ. Satellite cell content is specifically reduced in type II skeletal muscle fibers in the elderly. Am J Physiol Endocrinol Metab. 2007 Jan;292(1):E151-7. doi: 10.1152/ajpendo.00278.2006. Epub 2006 Aug 22. PMID 16926381
- [Result] Villacorta H, Bortolotto LA, Arteaga E, Mady C. Aortic distensibility measured by pulse-wave velocity is not modified in patients with Chagas' disease. J Negat Results Biomed. 2006 Jun 12;5:9. doi: 10.1186/1477-5751-5-9. PMID 16768804
- [Result] Wernbom, M. Effects of an acute bout of low-load resistance training with blood flow restriction. 2011. 206 f. Dissertation. The Norwegian School of Sports Sciences. Noruega. 2011.
- [Result] World Health Organization. Global brief for World Health Day. 2012. http://www.who.int/world_health_day/2012.
- [Result] Wu IC, Lin CC, Hsiung CA. Emerging roles of frailty and inflammaging in risk assessment of age-related chronic diseases in older adults: the intersection between aging biology and personalized medicine. Biomedicine (Taipei). 2015;5(1):1. doi: 10.7603/s40681-015-0001-1. Epub 2015 Feb 2. PMID 25722960
- [Result] Yasuda T, Loenneke JP, Thiebaud RS, Abe T. Effects of blood flow restricted low-intensity concentric or eccentric training on muscle size and strength. PLoS One. 2012;7(12):e52843. doi: 10.1371/journal.pone.0052843. Epub 2012 Dec 31. PMID 23300795
- [Result] Yasuda T, Fukumura K, Iida H, Nakajima T. Effects of detraining after blood flow-restricted low-load elastic band training on muscle size and arterial stiffness in older women. Springerplus. 2015 Jul 15;4:348. doi: 10.1186/s40064-015-1132-2. eCollection 2015. PMID 26191475
- [Result] Yasuda T, Fukumura K, Uchida Y, Koshi H, Iida H, Masamune K, Yamasoba T, Sato Y, Nakajima T. Effects of Low-Load, Elastic Band Resistance Training Combined With Blood Flow Restriction on Muscle Size and Arterial Stiffness in Older Adults. J Gerontol A Biol Sci Med Sci. 2015 Aug;70(8):950-8. doi: 10.1093/gerona/glu084. Epub 2014 Jun 10. PMID 24917178
- [Result] Yokokawa Y, Hongo M, Urayama H, Nishimura T, Kai I. Effects of low-intensity resistance exercise with vascular occlusion on physical function in healthy elderly people. Biosci Trends. 2008 Jun;2(3):117-23. PMID 20103914
- [Result] Nakajima, T.; Morita, T.; Sato, Y. Key considerations when conducting KAATSU training. International Journal of Kaatsu Training Research. 2011. v. 7. p. 1-6.
- [Derived] Amorim S, Degens H, Passos Gaspar A, De Matos LDNJ. The Effects of Resistance Exercise With Blood Flow Restriction on Flow-Mediated Dilation and Arterial Stiffness in Elderly People With Low Gait Speed: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Nov 1;8(11):e14691. doi: 10.2196/14691. PMID 31682588